CLINICAL TRIAL: NCT04417621
Title: A Randomized, Open-label, Multi-arm, Two-part, Phase II Study to Assess Efficacy and Safety of Multiple LXH254 Combinations in Patients With Previously Treated Unresectable or Metastatic BRAFV600 or NRAS Mutant Melanoma
Brief Title: Study of Efficacy and Safety of LXH254 Combinations in Patients With Previously Treated Unresectable or Metastatic Melanoma
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CLXH254C12201; 2020-000873-26 (EudraCT Number)
Record Dates: First submitted 2020-06-03; First posted 2020-06-04 (Actual); Last update posted 2025-10-21 (Actual); Status verified 2025-10

CONDITIONS: Melanoma
Keywords: LXH254; Melanoma; NRAS; BRAF; LTT462; Trametinib; Ribocliclib
MeSH Terms: conditions — Melanoma | interventions — naporafenib; trametinib; ribociclib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- LXH254 + LTT462 (Experimental)
  Interventions: Drug: LXH254; Drug: LTT462
- LXH254 + trametinib (Experimental)
  Interventions: Drug: Trametinib
- LXH254 + ribociclib (Experimental)
  Interventions: Drug: Ribociclib

INTERVENTIONS:
Drug: LXH254 — LXH254 will be supplied as tablet for oral use.
  Arms: LXH254 + LTT462
Drug: LTT462 — LTT462 will be supplied as hard gelatin capsule for oral use.
  Arms: LXH254 + LTT462
Drug: Trametinib — Trametinib will be supplied as film-coated tablet for oral use
  Arms: LXH254 + trametinib
Drug: Ribociclib — Ribociclib will be supplied in tablets and hard gelatin capsules.
  Arms: LXH254 + ribociclib

SUMMARY:
The primary purpose of this study is to evaluate the efficacy of LXH254 combinations in previously treated unresectable or metastatic melanoma

ELIGIBILITY:
Inclusion Criteria:

Male or female must be ≥ 12 years For adolescents only (12-17 years): body weight > 40kg Histologically confirmed unresectable or metastatic cutaneous melanoma

Previously treated for unresectable or metastatic melanoma:

* Participants with NRAS mutation:
* Participants must have received prior systemic therapy for unresectable or metastatic melanoma with checkpoint inhibitors (CPI), either an anti-PD-1/PD-L1 as a single agent or in combination with anti-CTLA-4, investigational agents, chemotherapy or locally directed anti-neoplastic agents.
* A maximum of two prior lines of systemic CPI-containing immunotherapy for unresectable or metastatic melanoma are allowed. Additional agents administered with CPI are permitted.
* To rule out pseudo-progression, participants must have documented confirmed progressive disease as per RECIST v1.1 while on/after treatment with checkpoint inhibitor therapy. Confirmation is not required for patients who remained on treatment for >6 months.
* Participants with BRAFV600 mutant disease:
* Participants must have received prior systemic therapy for unresectable or metastatic melanoma with checkpoint inhibitors (CPI), either an anti-PD-1/PD-L1 as a single agent or in combination with anti-CTLA-4, investigational agents, chemotherapy or locally directed anti-neoplastic agents. Additionally, participants must have received targeted therapy with a RAFi as a single agent or in combination with a MEKi (+/- CPI allowed) as the last prior therapy.
* A maximum of two prior lines of systemic CPI-containing immunotherapy for unresectable or metastatic melanoma are allowed. Additional agents with CPI are permitted.
* A maximum of one line of targeted therapy is allowed, and it must be the most recent line of therapy.
* Participants must have documented progressive disease as per RECIST v1.1 while on/after treatment with targeted therapy.

Other protocol-defined inclusion criteria may apply.

Exclusion Criteria:

Treatment with any of the following anti-cancer therapies prior to the first dose of study treatment within the stated timeframes:

* ≤ 4 weeks for radiation therapy or ≤ 2 weeks for limited field radiation for palliation prior to the first dose of study treatment.
* ≤ 2 weeks for small molecule therapeutics.
* ≤ 4 weeks for any immunotherapy treatment including immune checkpoint inhibitors.
* ≤ 4 weeks for chemotherapy agents, locally directed anti-neoplastic agents, or other investigational agents.
* ≤ 6 weeks for cytotoxic agents with major delayed toxicities, such as nitrosourea and mitomycin c.

Participants participating in additional parallel investigational drug or medical device studies.

All primary central nervous system (CNS) tumors or symptomatic CNS metastases that are neurologically unstable History or current evidence of retinal vein occlusion (RVO) or current risk factors for RVO (e.g. uncontrolled glaucoma or ocular hypertension, history of hyperviscosity or hypercoagulability syndromes).

Any medical condition that would, in the investigator's judgment, prevent the patient's participation in the clinical study due to safety concerns or compliance with clinical study procedures.

Other protocol-defined exclusion criteria may apply

Ages: 12 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 134 (Actual)
Dates: Start 2020-10-30 (Actual); Primary Completion 2026-03-27 (Estimated); Study Completion 2026-03-27 (Estimated)

PRIMARY OUTCOMES:
Overall Response Rate | 35 months
  Confirmed ORR using RECIST v1.1, per local assessment

SECONDARY OUTCOMES:
Duration of Reposnse (DOR) | 4 years
  Local and central assessment
Progression Free Survival (PFS) | 4 years
Disease Control Rate (DCR) | 3 years
  Using RECIST v1.1, per local and central assessment
Overall Survival (OS) | 4 years
Derived PK parameter (Cmax) for LXH254 & LTT462 | Up to 5 months
Derived PK parameter (Cmax) for LXH254 & trametinib | Up to 5 months
Derived PK parameter (Cmax) for LXH254 & ribociclib | Up to 5 months
Derived PK parameter (AUC) for LXH254 & LTT462 | Up to 5 months
Derived PK parameter (AUC) for LXH254 & trametinib | Up to 5 months
Derived PK parameter (AUC) for LXH254 & ribociclib | Up to 5 months
Incidence of adverse events (AEs) and serious adverse events (SAEs) | 35 months
  Number of participants with Adverse Events (AEs) and SAEs as a measure of safety and tolerability
Dose Interruptions | 35 months
  Tolerability measured by the number of subjects who have interruptions of study treatment and reason for interruptions
Dose reductions | 35 months
  Tolerability measured by the number of subjects who have reductions of study treatment and reason for reductions

CONTACTS AND LOCATIONS:
Locations (36):
- United States (12):
  - The Angeles Clinic and Research Institute, Los Angeles, California
  - UCSF Medical Center, San Francisco, California
  - Florida Cancer Specialists, Fort Myers, Florida
  - H Lee Moffitt Cancer Center and Research Institute, Tampa, Florida
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Mayo Clinic Mayo Rochester, Rochester, Minnesota
  - Mayo Clinic Rochester, Rochester, Minnesota
  - NYU Laura and Isaac Perlmutter Cancer Center, New York, New York
  - Memorial Sloan Kettering, New York, New York
  - University of Pittsburgh Med Center, Pittsburgh, Pennsylvania
  - Univ of TX MD Anderson Cancer Cntr, Houston, Texas
- Novartis Investigative Site, CABA, Buenos Aires, Argentina
- Australia (3):
  - Novartis Investigative Site, North Sydney, New South Wales
  - Novartis Investigative Site, Wooloongabba, Queensland
  - Novartis Investigative Site, Subiaco, Western Australia
- Belgium (2):
  - Novartis Investigative Site, Leuven
  - Novartis Investigative Site, Wilrijk
- France (6):
  - Novartis Investigative Site, Lille
  - Novartis Investigative Site, Marseille
  - Novartis Investigative Site, Paris
  - Novartis Investigative Site, Pierre-Bénite
  - Novartis Investigative Site, Toulouse
  - Novartis Investigative Site, Villejuif
- Germany (4):
  - Novartis Investigative Site, Dresden, Saxony
  - Novartis Investigative Site, Essen
  - Novartis Investigative Site, Heidelberg
  - Novartis Investigative Site, Tübingen
- Novartis Investigative Site, Ramat Gan, Israel
- Italy (2):
  - Novartis Investigative Site, Milan, MI
  - Novartis Investigative Site, Napoli
- Novartis Investigative Site, Maastricht, Limburg, Netherlands
- Novartis Investigative Site, Oslo, Norway
- Switzerland (2):
  - Novartis Investigative Site, Lausanne
  - Novartis Investigative Site, Zurich
- Novartis Investigative Site, Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations. This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com.

REFERENCES:
- [Derived] Moschos SJ. War against NRAS-Mutant Melanoma Using Targeted Therapies Remains Challenging. Clin Cancer Res. 2022 Jul 15;28(14):2977-2979. doi: 10.1158/1078-0432.CCR-22-1256. PMID 35587446